CLINICAL TRIAL: NCT06348485
Title: Massive Nasal Bleeding in Patients With Nasopharyngeal Carcinoma Received Curative Radiotherapy
Brief Title: Massive Nasal Bleeding in Patients With NPC Received Curative RT
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Hao-Shen Cheng, Attending Physician, Taichung Veterans General Hospital
Other Study IDs: VGHTCCTC_NPCbleeding001
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma Patients Treated With Curative Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NPC received Curative radiotherapy
  Interventions: Other: Patients without massive nasal bleeding; Other: Patients with massive nasal bleeding

INTERVENTIONS:
Other: Patients without massive nasal bleeding — No event of massive nasal bleeding after curative radiotherapy
Other: Patients with massive nasal bleeding — Any event of massive nasal bleeding after curative radiotherapy

SUMMARY:
To investigate the incidence, predictive markers, and survival impact of massive nasal bleeding in nasopharyngeal carcinoma (NPC) patients who received curative radiotherapy (RT) with/without chemotherapy. A total of 1327 patients with previously untreated, biopsy-proven NPC, and no distant metastasis were retrospective reviewed. Investigators analyzed the occurrence rates of massive nasal bleeding between different characteristics and tried to identify important predictive factors. Investigators compared overall survival between patients with and without massive nasal bleeding by Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* previously untreated, biopsy-proven NPC
* no distant metastasis

Exclusion Criteria:

* incomplete record of history or treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1327 patients with previously untreated, biopsy-proven NPC, and no distant metastasis were retrospective reviewed. There are 957 males and 370 females received conventional 2D or 3D conformal radiotherapy.
Sampling Method: Probability Sample
Enrollment: 1327 (Actual)
Dates: Start 1994-12-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Massive Nasal Bleeding Rate | From date of radiotherapy until the date of first documented massive bleeding, assessed up to 360 months
  Massive Nasal Bleeding Rate among different characteristics. Massive Nasal Bleeding was defined as unique blood loss > 300 ml or recurrent blood losses > 100 ml.

SECONDARY OUTCOMES:
Overall Survival | From date of radiotherapy until the date of last clinic visit or date of death from any cause, whichever came first, assessed up to 360 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang Y, Yan D, Wang M, Chen S, Yang F. Clinicopathological factors affecting the prognosis of massive hemorrhage after radiotherapy for patients having nasopharyngeal carcinoma. J Cancer Res Ther. 2021 Nov;17(5):1219-1224. doi: 10.4103/jcrt.jcrt_586_21. PMID 34850770
- [Background] Zhan J, Zhang S, Wei X, Fu Y, Zheng J. Etiology and management of nasopharyngeal hemorrhage after radiotherapy for nasopharyngeal carcinoma. Cancer Manag Res. 2019 Mar 15;11:2171-2178. doi: 10.2147/CMAR.S183537. eCollection 2019. PMID 30936749
- [Background] Li J, Yi X, He G, Yao D, Bin X, Feng Y, Niu Z, Tan Q, Tang A. Analysis of the risk of death and clinical management for nasal or nasopharyngeal bleeding occurring after radiotherapy for nasopharyngeal carcinoma. Auris Nasus Larynx. 2022 Aug;49(4):703-708. doi: 10.1016/j.anl.2022.01.006. Epub 2022 Jan 20. PMID 35065845
- [Background] Zeng L, Wan W, Luo Q, Jiang H, Ye J. Retrospective analysis of massive epistaxis and pseudoaneurysms in nasopharyngeal carcinoma after radiotherapy. Eur Arch Otorhinolaryngol. 2022 Jun;279(6):2973-2980. doi: 10.1007/s00405-021-07111-x. Epub 2021 Oct 8. PMID 34623497